CLINICAL TRIAL: NCT00096499
Title: A Phase II Study of SB-715992 (NSC-727990, IND-70273) in Taxane-Resistant Androgen-Independent Metastatic Prostate Cancer
Brief Title: SB-715992 in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Docetaxel or Paclitaxel
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02630; SWOG-S0418; U10CA032102 (NIH); CDR0000393206 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-11-09; First posted 2004-11-10 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ispinesib; CK0238273

ARMS (1):
- Treatment (ispinesib) (Experimental): Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ispinesib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ispinesib — Given IV
  Other Names: CK0238273; SB-715992
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as SB-715992, work in different ways to stop tumor cells from dividing so they stop growing or die. This phase II trial is studying how well SB-715992 works in treating patients with metastatic prostate cancer that did not respond to docetaxel or paclitaxel

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the prostate-specific antigen response to SB-715992 in patients with hormone-refractory, androgen-independent metastatic prostate cancer that failed prior taxane-based chemotherapy.

SECONDARY OBJECTIVES:

I. Determine the median overall survival and median progression-free survival of patients treated with this drug.

II. Determine the objective response rate (confirmed and unconfirmed, complete and partial response) in patients with measurable disease treated with this drug.

III. Determine the qualitative and quantitative toxic effects of this drug in these patients.

IV. Determine, preliminarily, the pharmacokinetics and mechanism of activity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive SB-715992 IV over 1 hour on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 1.3-2.7 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic disease (N1 and/or M1)
  * Unresponsive or refractory to androgen-deprivation therapy
* Must have received one, and only one, prior taxane-containing (docetaxel or paclitaxel) chemotherapy regimen for metastatic disease that was discontinued due to disease progression, intolerance, or patient request
* Evidence of disease progression as defined by ≥ 1 of the following:

  * Progression of measurable disease
  * Progression of evaluable disease
  * Rising prostate-specific antigen (PSA)

    * At least 2 consecutive rises in PSA levels, each taken ≥ 7 days apart
    * PSA ≥ 5 ng/mL
* Must have pre-study PSA > 5 ng/mL
* Measurable or evaluable disease

  * Soft tissue disease that has been irradiated within the past 2 months is not considered measurable disease
  * Soft tissue disease that has been irradiated ≥ 2 months prior to study entry is considered measurable disease provided the lesion progressed after radiation
* Surgical or medical castration required

  * If luteinizing hormone-releasing hormone (LHRH) agonists (leuprolide or goserelin) or LHRH antagonists (abarelix) were used, then must continue use during study therapy
* No prior or concurrent brain metastases (treated or untreated)

  * If clinical suspicion of brain metastases, must meet the following criteria:

    * Brain CT scan or MRI negative for metastatic disease within the past 56 days
    * No new symptoms since radiographic evaluation
* Performance status - Zubrod 0-2
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Bilirubin normal
* SGOT and SGPT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance ≥ 40 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Fertile patients must use effective contraception
* No peripheral neuropathy ≥ grade 2
* No prior allergic reaction attributed to compounds of similar chemical or biological composition to SB-715992
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation
* No other uncontrolled illness
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated stage I or II cancer in complete remission
* No colony-stimulating factors during the first course of study therapy
* No concurrent anticancer biologic therapy
* See Disease Characteristics
* At least 4 weeks since prior chemotherapy and recovered
* See Disease Characteristics
* At least 4 weeks since prior flutamide or ketoconazole
* At least 6 weeks since prior bicalutamide or nilutamide
* No concurrent anticancer hormonal therapy except LHRH agonist or antagonist for patients who have not undergone orchiectomy
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy and recovered
* Prior samarium Sm 153 lexidronam pentasodium allowed
* No prior strontium chloride Sr 89
* No prior radiotherapy to ≥ 30% of bone marrow
* No concurrent anticancer radiotherapy
* See Disease Characteristics
* At least 3 weeks since prior surgery and recovered
* At least 2 weeks since prior and no concurrent use of any of the following CYP3A4 inhibitors or inducers:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Rifampin
  * Rifabutin
  * Rifapentine
  * Itraconazole
  * Ketoconazole
  * Fluconazole (dose > 200 mg/day)
  * Voriconazole
  * Nefazodone
  * Fluvoxamine
  * Verapamil
  * Diltiazem
  * Grapefruit juice
  * Bitter orange
  * Phenytoin
  * Carbamazepine
  * Phenobarbital
  * Oxcarbazepine
  * Hypericum perforatum (St. John's wort)
  * Modafinil
* At least 6 months since prior and no concurrent amiodarone
* No other investigational drugs for 4 weeks before, during, and for 2 weeks after study therapy
* No other concurrent anticancer cytotoxic therapy
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* Concurrent enrollment on SWOG-9205 (central prostate cancer serum repository protocol) allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-04; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Probability of PSA response | Up to 3 years

SECONDARY OUTCOMES:
Overall survival | From date of registration to date of death due to any cause, assessed up to 3 years
Progression-free survival | From date of registration to date of first observation of progressive disease, symptomatic deterioration, or death due to any cause, assessed up to 3 years
Probability of objective response | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Beer, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States